CLINICAL TRIAL: NCT02731521
Title: Clinical Development of MR Spectroscopy and Imaging in Brain Cancers
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Sponsor
Other Study IDs: STU 122013-077
Record Dates: First submitted 2016-03-02; First posted 2016-04-07 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Malignant Gliomas; Astrocytomas; Oligodendrogliomas
Keywords: MRS Biomarkers
MeSH Terms: conditions — Glioma; Astrocytoma; Oligodendroglioma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 3 Tesla Scanning and 7 Tesla Scanning: Scanning at 3 Tesla and 7 Tesla: Magnetic Resonance Imaging (MRI)/Magnetic Resonance Spectroscopy (MRS) of glioma and non-glioma patients.
  Interventions: Device: 3 Tesla Scanning; Device: 7 Tesla Scanning

INTERVENTIONS:
Device: 3 Tesla Scanning — Approximately 120 brain tumor patients 50 patients with non-glioma disease, and 5 healthy volunteers will be scanned at either 3 Tesla or 7 Tesla.
  Other Names: 3T MRI/MRS
Device: 7 Tesla Scanning — Approximately 120 brain tumor patients 50 patients with non-glioma disease, and 5 healthy volunteers will be scanned at either 3 Tesla or 7 Tesla.
  Other Names: 7T MRI/MRS

SUMMARY:
The Investigators will examine the disease specificity of 2-hydroxyglutarate in non-glioma brain lesions, and the clinical utility of 2-hydroxyglutarate, glycine and citrate in isocitrate dehydrogenase (IDH) mutated gliomas and IDH wild type gliomas.

DETAILED DESCRIPTION:
2-hydroxyglutarate (2HG) imaging will identify glioma, tumor progression and response to therapy noninvasively at an earlier time point than currently detectable with standard MR imaging. This utility of 2HG can be used for improving the patient care in a more effective manner when the 2HG imaging is incorporated in regular clinical MR scans in brain tumor patients. We aim to translate the 2HG MRS protocol into two clinical MR centers at UTSouthwestern Medical Center: The Mary Nell and Ralph B. Rogers Magnetic Resonance Center with Philips 1.5Tesla and 3Tesla scanners and The Algur H. Meadows Diagnostic Imaging Center with a GE 3Tesla scanner. In addition, we will perform Magnetic Resonance (MR) scans in patients with neurological diseases that can mimic gliomas, including stroke, epilepsy, encephalitis, and brain metastases in order to establish the specificity of 2HG to malignant gliomas.

ELIGIBILITY:
Inclusion Criteria:

(120 Brain Tumor Patients)

* All races and ethnicities
* Must meet at least one of the 3 following criteria regarding diagnosis:

  * Histological diagnosis of a brain tumor
  * Pre-operative MR imaging suggestive of a brain tumor
  * Radiographic diagnosis of brain tumor in an inoperable location (e.g. brainstem)
* Pretreatment evaluations required for eligibility include a medical history, physical examination, and neurological exam within 30 days prior to study entry.
* Patient must be able to provide study-specific consent prior to study entry and Health Insurance Portability and Accountability Act of 1996 (HIPAA) authorization.
* Karnofsky performance status >70%
* Life expectancy greater than 3 months.

  (50 Non-Tumor Neurological Disorders)
* All races and ethnicities
* Patients with clinically-proven multiple sclerosis, temporal lobe epilepsy, stroke, or encephalitis.

  (5 Health Volunteers)
* 18-40 years of age
* All races and ethnicities
* Excellent general health

Exclusion Criteria:

* Under age 18
* Cardiac pacemaker
* Intracranial clips, metal implants, or external clips within 50 cm from the head
* Metal in eye
* Pregnancy
* Claustrophobia
* Obesity or any other factors that provide difficulty with supine pose in the magnet
* Patients who are unable to provide informed consent
* Patients who are pregnant or nursing
* Patients with severe kidney dysfunction or uncontrolled cardiac dysfunction
* Patients who are claustrophobic or have other contraindication to MRI, such as implanted pacemaker device, vascular clips, surgical clips, prosthetic valves, pace¬makers, otologic implants
* Patients with uncontrolled psychiatric manifestations of their brain tumor
* Patients for 7 Tesla scans can have no metal in the body

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Glioma patients recruited from UTSW neurosurgery and neuro-oncology clinics.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2014-01; Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Amount of 2-hydroxyglutarate (2HG) bio-marker in 170 patients with clinically-proven brain metastasis, multiple sclerosis, epilepsy, stroke, or encephalitis using magnetic resonance spectroscopy (MRS). | 1-4 scans, average over 36 months
  Measuring amount of 2-hydroxygluterate (2HG) biomarker with MRS.

CONTACTS AND LOCATIONS:
Overall Officials: Changho Choi, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided